CLINICAL TRIAL: NCT06205069
Title: The Immediate Effects of Tissue Flossing on Knee Flexion Range of Motion: A Randomized Controlled Trial
Brief Title: The Immediate Effects of Tissue Flossing on Knee Flexion Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Principal Investigator, Ricardo Cardoso, Professor, University Fernando Pessoa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ESS/FSA - 320/22
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The floss band will be applied to the knee of the dominant lower limb in the intervention group (IG). While the participant will stand and perform a slight knee flexion, the band will be rolled upwards from the tibial tuberosity to 5 cm above the femoral epicondyle. The patella will not be covered. Pressure will be produced by rolling the joint with 50% tension and 50% overlap.
  After applying the floss band, passive mobilization will be performed - 20 repetitions of knee flexion and extension and an active movement task - 20 squats. Participants will be instructed to perform knee flexion and extension to their extreme range of motion and to complete the mobility exercises within two minutes. After two minutes, the floss band will be removed and participants will be instructed to stand up and walk for a minute to allow blood to flow back to the foot.
  Interventions: Device: Tissue flossing
- Control group (No Intervention): For the CG, after initial assessment, participants without a floss band will perform the same two functional movement tasks (active and passive) with 20 repetitions as the GI for 2 minutes. After two minutes, participants will be instructed to get up and walk for one minute like the intervention group.

INTERVENTIONS:
Device: Tissue flossing — While the participant will stand and perform a slight knee flexion, the band will be rolled upwards from the tibial tuberosity to 5 cm above the femoral epicondyle. The patella will not be covered. Pressure will be produced by rolling the joint with 50% tension and 50% overlap.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to verify the immediate effects of Tissue Flossing on knee flexion range of motion

DETAILED DESCRIPTION:
After completing the questionnaire, 58 healthy participants will be randomly divided into two groups named Intervention Group (IG) (n=29) and Control Group (CG) (n=29).

In the first assessment (M0), knee flexion ranges will be measured using a goniometer. Then the control group (n=29), without Tissue Flossing and intervention group (n=29) with Tissue Flossing around the knee joint will be subjected to passive and then active mobilization of the knee joint. Immediately after the intervention/control, the two groups will be assessed again (M1).

ELIGIBILITY:
Inclusion Criteria:

* healthy people between 18 and 35 years old with normal mobility of the joints of the lower limbs of the body.

Exclusion Criteria:

* deformities in the region of the lower limbs of the body, complaints in this region in the last 6 months, surgical procedures, venous thrombotic disease, heart disease, respiratory disease, or neurological, orthopedic, dermatitis, or neuromuscular problems in the lower quadrant that may disrupt musculoskeletal function. Also high blood pressure, latex allergies, lymphedema and individuals taking anticoagulant medication, and cortisteroid therapy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Change of knee range of motion | [Time Frame: Change from Baseline (M0) to Immediately after intervention or control (M1)]
  Data will be collected in two moments: baseline (M0) and after the intervention/control (M1).
  The knee flexion range of motion will be measured using a smartphone app "Goniometer Pro". The distance between the lateral femoral epicondyle and the center of the lateral malleolus will be assessed. To measure the knee flexion angle, the participant will be placed in the prone position with the hip and knee extended at 0° (goniometer initial position 0°) with the foot relaxed and the contralateral leg extended. For active range of motion, the participant will be asked to perform maximum knee flexion in the prone position. To measure passive movement, the examiner will perform maximum knee flexion on participants in the same position. The average of three repetitions of ranges of movement will be recorded with 30-second rest intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior Saúde Fernando Pessoa, Porto, Portugal